CLINICAL TRIAL: NCT03491839
Title: A Modeling of Changes in Tidal Volume With Concentration of Inhalational Anesthetics Under General Anesthesia Using Laryngeal Mask Airway
Brief Title: A Modeling of Changes in Tidal Volume With Concentration of Inhalational Anesthetics
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, professor, Seoul National University Hospital
Other Study IDs: 1803-068-929
Record Dates: First submitted 2018-04-01; First posted 2018-04-09 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
modelling of tidal volume with inhalational anesthetic concentration

DETAILED DESCRIPTION:
The investigators would like to develop the modelling of tidal volume with inhalational anesthetic concentration during spontaneous breathing during general anesthesia in children

ELIGIBILITY:
Inclusion Criteria:

- general anesthesia

Exclusion Criteria:

-

Max Age: 12 Years | Sex: All
Age Groups: Child
Study Population: children under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
concentration | 20 minutes
  inhalational anesthetic concentration

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea